CLINICAL TRIAL: NCT07010055
Title: Using Digital Health in a Postoperative Setting After Major Surgery: a Prospective Single-center Qualitative Semi-structured Interview Study
Brief Title: Using Digital Health in a Postoperative Setting After Major Surgery: Semi-structured Interview Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Professor, Dr, Jessa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/046
Record Dates: First submitted 2025-05-27; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Digital Health
Keywords: Remote monitoring; Major surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-structured interview (Experimental): Conducting a semi-structured interview during a follow-up consultation after major surgery
  Interventions: Procedure: Semi-structured interview

INTERVENTIONS:
Procedure: Semi-structured interview — A semi-structured interview will be conducted once in-person to each patient after a follow-up consultation in the hospital after their major surgery

SUMMARY:
This study aims to evaluate whether patients recognize a need for a remote monitoring care pathway during the post-operative period following major surgery at Jessa Hospital by means of a semi- structured interview. Besides this, the study explores patient perceptions and willingness to participate in digital monitoring care pathways, identifies potential barriers to adoption, and addressing concerns related to safety, data security, and privacy. Additionally, the study aims to assess patient needs regarding parameter collection, technology usage, and the overall functionality of digital monitoring systems, while evaluating the perceived usefulness of such a pathway in post-operative care.

DETAILED DESCRIPTION:
Digital health technologies are transforming healthcare, offering new ways to improve patient outcomes and enhance efficiency. Remote clinical monitoring (RCM), which uses digital technologies such as wearable devices and mobile apps to monitor patients outside of the traditional healthcare settings such as a hospital, holds significant potential for supporting post-operative care, especially in the context of faster hospital discharge after major surgery. Major surgery involves procedures on organ systems, such as cancer resections, organ transplants, and lung or abdominal surgeries. However, despite their promise, the successful implementation of these technologies into clinical practice requires a thorough understanding of the perspectives of the end user, being the patient. Patients' comfort, engagement, and perceptions about digital health solutions, such as self-management tools and remote monitoring pathways, are essential to ensuring these technologies are both effective and widely accepted.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients

  * >18 years old, Undergone major surgery at Jessa Hospital Hasselt

Exclusion Criteria:

* Unable to provide informed consent or request to not participate in the study
* Cognitively incapable of understanding the study
* No understanding of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Need for monitoring of vital and subjective parameters after discharge | During a follow-up consultation within one year after major surgery
  The primary outcome measurement will be assessed by asking patients if they believe that there is a need for monitoring of vital and subjective parameters after discharge.

SECONDARY OUTCOMES:
Perceptions regarding the implementation of digital monitoring care pathways | During a follow-up consultation within one year after major surgery
  Patients' perceptions regarding the implementation of digital monitoring care pathways will be evaluated by asking questions about their experience and knowledge of remote care, their perceptions of whether digital monitoring can replace traditional face-to-face consultations, their need for digital information after discharge, and their experience with follow-up and contact with healthcare providers after discharge.
Willingness to participate in digital care pathways | During a follow-up consultation within one year after major surgery
  To examine patients' willingness to participate in digital care pathways, following items are questioned: willingness to be discharged sooner with remote monitoring available, factors that would motivate patients to use or recommend remote monitoring, and comfort and willingness to have health monitored remotely through an app or device.
Potential barriers to adopt digital care | During a follow-up consultation within one year after major surgery
  To identify potential barriers to adopt digital care, challenges in using remote care will be surveyed.
Concerns about safety | During a follow-up consultation within one year after major surgery
  Patients' concerns about safety when being discharged earlier with remote monitoring in place are assessed to understand patient concerns about their own safety.
Accuracy of data | During a follow-up consultation within one year after major surgery
  Trust in the accuracy of data collected through remote monitoring and security of personal data when using remote monitoring are evaluated to understand patient concerns regarding data security and privacy.
Needs regarding parameter collection | During a follow-up consultation within one year after major surgery
  To understand patient needs regarding parameter collection, patients are asked if they think there is a need for additional parameters to be collected beyond vital signs (e.g., blood pressure, oxygen saturation, body temperature, heart rate), or if they have specific preferences for health parameters to be collected.
Skills regarding working with technology | During a follow-up consultation within one year after major surgery
  To examine patients' skills regarding working with technology, skills in using technology, comfort using digital devices for health monitoring, and the need for training to use remote monitoring effectively will be investigated.
Desire for notifications when a parameter or questionnaire needs to be entered in an app | During a follow-up consultation within one year after major surgery
  The desire for notifications when a parameter or questionnaire needs to be entered in an app, for alerts or alarms when a parameter is abnormal, for digital feedback from healthcare providers, or to communicate directly with healthcare providers through an app is explored to understand patient needs regarding the functioning of the digital monitoring care pathway.
Perceptions regarding the usefulness of a digital monitoring care pathway | During a follow-up consultation within one year after major surgery
  To assess patient perceptions regarding the usefulness of a digital monitoring care pathway, their perception of the potential for remote monitoring to improve the recovery process, of benefits for patients/healthcare providers/society, of remote monitoring helping to reduce anxiety about recovery through continuous monitoring, and of remote monitoring helping to prevent complications, will be examined.
Willingness to participate in a study with remote monitoring | During a follow-up consultation within one year after major surgery
  The willingness to participate in a study with remote monitoring is asked to assess patient willingness to participate in a study where digital monitoring is used.